CLINICAL TRIAL: NCT04962945
Title: Comparison of the Oblique-axis and Long-axis Approaches for Axillary Vein Catheterization Under Ultrasound Guidance in Cardiac Surgery Patients Susceptible to Bleeding: a Randomized Controlled Trial
Brief Title: Comparison of the Oblique-axis and Long-axis Approaches for Axillary Vein Catheterization Under Ultrasound Guidance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guowei Tu (Other)
Responsible Party: Sponsor-Investigator, Guowei Tu, Scientific Secretary for Department of Critical Care Medcine, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2021-018R
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Central Venous Catheterization
Keywords: axillary vein; central venous catheterization; ultrasound; cardiac surgery; complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oblique-axis approach group (Active Comparator): The first two attempts via the oblique-axis approach will be performed . If the first two attempts failed, the subsequent attempts of venipuncture were performed using the long-axis approach.
  Interventions: Procedure: Oblique-axis approach group
- Long-axis approach group (Active Comparator): The first two attempts via the long-axis approach will be performed . If the first two attempts failed, the subsequent attempts of venipuncture were performed using the oblique-axis approach.
  Interventions: Procedure: Long-axis approach group

INTERVENTIONS:
Procedure: Oblique-axis approach group — The first two attempts via the oblique-axis approach will be performed . If the first two attempts failed, the subsequent attempts of venipuncture were performed using the long-axis approach.
  Arms: Oblique-axis approach group
Procedure: Long-axis approach group — The first two attempts via the long-axis approach will be performed . If the first two attempts failed, the subsequent attempts of venipuncture were performed using the oblique-axis approach.
  Arms: Long-axis approach group

SUMMARY:
Ultrasound-guided axillary vein catheterization can be performed via the oblique-axis and long-axis approaches of the axillary vein. The aim of our study is to compare the first puncture success rate and safety between the two approaches of ultrasound-guided axillary vein catheterization in cardiac surgical patients with high bleeding risk

DETAILED DESCRIPTION:
For patients after cardiac surgery, antiplatelet drugs or anticoagulants are usually used for preventing thrombosis. Use of those drugs is associated with increased risk of bleeding. Any invasive procedures may put those patients at additional risk of bleeding. Ultrasound (US) has become widely accepted to guide safe and accurate central venous catheterization. Ultrasound-guided axillary vein catheterization can be performed via the oblique-axis and long-axis approaches of the axillary vein. The aim of our study is to compare the first puncture success rate and safety between the two approaches of ultrasound-guided axillary vein catheterization in cardiac surgical patients with high bleeding risk

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgical patients in Cardiac Surgery Intensive Care Unit
* Axillary vein catheterization is needed according to the clinical practice

Exclusion Criteria:

* the proximal and/or distal axillary vein was not clearly visualized or potentially unavailable for catheterization;
* did not receive or had not received oral antiplatelet drugs and/or anticoagulants for less than 3 days;
* already had presence of subclavian or axillary vein catheter;
* required an emergency axillary vein catheterization;
* had fracture of the ipsilateral clavicle or anterior proximal ribs;
* had subclavian and/or axillary vein thrombosis;
* had local infection of the puncture area.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
First puncture success rate | approximately 3-5 minutes
  Central venous catheter established upon first punction attempt

SECONDARY OUTCOMES:
approach success rate | within 1 hours
  the number of successful cannulation within the first two attempts
strategy success rate | within 1 hours
  defined as the number of successful cannulation in targeted axillary vein within four attempts (the first two attempts using the randomized approach, third and fourth attempts using the non-randomized approach)
the number of attempts | within 1 hours
  the number of attempts until successful cannulation
access time | within 1 hours
  defined as the time between penetration of skin and aspiration of venous blood into the syringe
time to successful cannulation | within 1 hours
  the time from skin puncture until completion of cannula insertion
Complications rate | 1 day
  Complications included arterial puncture, pneumothorax, haemothorax, nerve injuries, hematoma, catheter misplacement

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, Professor, Study Director — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided